CLINICAL TRIAL: NCT00506935
Title: Phase 1 Study of Vigabatrin (GVG) for Methamphetamine Dependence
Brief Title: Assessment of GVG for the Treatment of Methamphetamine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Thomas Newton, Professor, Baylor College of Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: #05-10-091-01
Record Dates: First submitted 2007-07-24; First posted 2007-07-25 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Methamphetamine Addiction
Keywords: methamphetamine; GVG; vigabatrin; stimulant
MeSH Terms: interventions — Vigabatrin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): GVG
  Interventions: Drug: GVG
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: GVG — 5 grams GVG
  Other Names: vigabatrin
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
The purpose of this study is to find out if GVG can reduce drug use and determine safety and effects of GVG when used together with methamphetamine. This study involves staying in the hospital for 21 days. Participants will receive either placebo or GVG, and a limited amount if methamphetamine will be injected on some study days. This study will enroll people that use methamphetamine. Participants will be compensated.

ELIGIBILITY:
Inclusion Criteria:

1. Be English-speaking volunteers who are not seeking treatment at the time of the study;
2. Be between 18-55 years of age;
3. Meet DSM-IV TR criteria for MA abuse or dependence;
4. Have a self-reported history of using MA by the smoked or IV route, for at least 2 years.
5. Have vital signs as follows: resting pulse between 50 and 90 bpm, blood pressures between 85-150mm Hg systolic and 45-90mm Hg diastolic; this criterion must be met within 2 days of admission.
6. Have hematology and chemistry laboratory tests that are within normal (+/- 10%) limits with the following exceptions: a) liver function tests (total bilirubin, ALT, AST, and alkaline phosphatase) < 3 x the upper limit of normal, and b) kidney function tests (creatinine and BUN) < 2 x the upper limit of normal;
7. Have a baseline ECG that demonstrates normal sinus rhythm, normal conduction, and no clinically significant arrhythmias;
8. Be able to fully cooperate with visual field testing to the point that a valid test is obtained during screening/baseline.
9. In the judgment of the study ophthalmologist, have visual fields within normal limits for age during the screening/baseline measurements;
10. Have acceptable ERG results for initiation of treatment with GVG (in the judgment of Drs. Nusinowitz and Newton, with ophthalmologic consultation as needed) , including having a value of the 30 Hz Flicker a-b amplitude as measured during the screening/baseline electroretinogram evaluations of 52 μV or above;
11. Have a medical history and brief physical examination demonstrating no clinically significant contraindications for study participation, in the judgment of the admitting physician and the principal investigator.

Exclusion Criteria:

1. Have any history or evidence suggestive of seizure disorder or brain injury;
2. Have any previous medically adverse reaction to MA, including loss of consciousness, chest pain, or epileptic seizure;
3. Have neurological or psychiatric disorders, such as:

   * psychosis, bipolar illness or major depression as assessed by the MINI;
   * organic brain disease or dementia assessed by clinical interview;
   * history of any psychiatric disorder which would require ongoing treatment or which would make study compliance difficult;
   * history of suicide attempts within the past three months assessed by the MINI and/or current suicidal ideation/plan as assessed by the MINI;
4. Have evidence of clinically significant heart disease or hypertension, as determined by the PI;
5. Have a family history in first-degree relatives of early cardiovascular morbidity or mortality, as determined by the PI;
6. Have any ophthalmologic disorder (e.g., glaucoma, cataracts, optic nerve disease, fixation problems, etc.) which, in the judgment of the study ophthalmologist, would:

   * make it difficult to obtain valid ophthalmologic perimetry, or electroretinography (ERG) assessments, or
   * increase the risks of visual side effects associated with VGB.
7. Have evidence of untreated or unstable medical illness including: neuroendocrine, autoimmune, renal, hepatic, or active infectious disease;
8. Have HIV and are currently symptomatic, have a diagnosis of AIDS, or are receiving antiretroviral medication;
9. Be pregnant or nursing. Other females must either be unable to conceive (i.e., surgically sterilized, sterile, or post-menopausal) or be using a reliable form of contraception (e.g., abstinence, birth control pills, intrauterine device, condoms, or spermicide). All females must provide negative pregnancy urine tests before study entry, upon hospital admission, and at the end of study participation;
10. Have any history of asthma, chronic coughing and wheezing, or other respiratory illnesses;
11. Currently use alpha or beta agonists, theophylline, or other sympathomimetics;
12. Have any other illness, condition, or use of medications, which in the opinion of the PI and/or the admitting physician would preclude safe and/or successful completion of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2006-07; Primary Completion 2008-04 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States